CLINICAL TRIAL: NCT06133920
Title: Immobilization Versus Early Range of Motion in Reverse Total Arthroplasty in Patients With Proximal Humerus Fractures
Brief Title: Duration of Immobilization After Reverse Total Arthroplasty for Proximal Humerus Fractures
Status: Recruiting | Type: Observational
Sponsor: The Cooper Health System (Other)
Responsible Party: Principal Investigator, Catherine Fedorka MD, Orthopaedic Surgeon, Assistant Professor of Orthopaedic Surgery, Assistant Program Director, Orthopaedic Surgery Residency Program, The Cooper Health System
Other Study IDs: IRB #20-533
Record Dates: First submitted 2023-07-26; First posted 2023-11-18 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Proximal Humeral Fracture; Reverse Total Shoulder Arthroplasty
Keywords: Proximal Humerus Fracture; Range of Motion; Immobilization
MeSH Terms: conditions — Shoulder Fractures | interventions — Immobilization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immobilization Group: The immobilization group will be placed in a shoulder abduction sling immediately after surgery for four weeks. They will be allowed to start gentle passive range of motion with forward flexion to 120 degrees, abduction to 90 degrees, and external rotation to 30 degrees. They will receive a home exercise program and formal physical therapy with these limits.
  When they come out of the sling at four weeks they will start active range of motion and active assisted range of motion. They cannot internally rotate until 10 weeks after surgery. No formal strengthening until 3 months after surgery.
  Interventions: Other: Immobilization
- Early ROM: The early range of motion group will be given a sling for comfort after their surgery. They will be told they can use their arm as tolerated and can remove the sling when comfortable immediately after surgery. They will be allowed to start passive range of motion, active assisted range of motion, and gentle active range of motion with therapy as tolerated with the exception of no internal rotation. They will also not be allowed to strengthen until 12 weeks after surgery. They will get formal physical therapy and be given a home exercise program as well that will be directed by their physical therapist
  Interventions: Other: Early Range of Motion

INTERVENTIONS:
Other: Early Range of Motion — The early range of motion group will be given a sling for comfort after their surgery. They will be told they can use their arm as tolerated and can remove the sling when comfortable immediately after surgery. They will be allowed to start passive range of motion, active assisted range of motion, and gentle active range of motion with therapy as tolerated with the exception of no internal rotation. They will also not be allowed to strengthen until 12 weeks after surgery. They will get formal physical therapy and be given a home exercise program as well that will be directed by their physical therapist
  Groups: Early ROM
Other: Immobilization — The immobilization group will be placed in a shoulder abduction sling immediately after surgery for four weeks. They will be allowed to start gentle passive range of motion with forward flexion to 120 degrees, abduction to 90 degrees, and external rotation to 30 degrees. They will receive a home exercise program and formal physical therapy with these limits.
  When they come out of the sling at four weeks they will start active range of motion and active assisted range of motion. They cannot internally rotate until 10 weeks after surgery. No formal strengthening until 3 months after surgery.
  Groups: Immobilization Group

SUMMARY:
The purpose of this study is to evaluate compare postoperative range of motion in patients who are given a sling for comfort only and allowed to start early active range of motion compared to patients who are placed in a sling for 4 weeks with passive range of motion only. Once enrolled, the patients will be randomized through computer randomization then placed in paper packets into either the immobilization group or the early range of motion group.

DETAILED DESCRIPTION:
Reverse shoulder arthroplasty is often used for older patients with displaced proximal humerus fractures in the older patient population. Many surgeons have historically placed patients in a sling for 4-6 weeks after surgery to prevent dislocation or tuberosity displacement. More recently though, surgeons are becoming more lenient with these restrictions as they realize it is very difficult for an elderly patient to be immobilized for 4-6 weeks. There has been one randomized control trial looking at early range of motion versus immobilization for 6 weeks after a regular reverse total shoulder arthroplasty not done for fracture which showed no difference at one year. There have not been any studies to date looking at reverse total shoulder arthroplasty for fracture to see if there is any difference in range of motion at early or later time points and also if there is an increased risk of complications.

Preoperative visit/hospitalization: The patient will be identified as meeting inclusion criteria and the study will be explained to them. Patients will be given a consent form to review with adequate time to review and decide if they wish to participate. If they choose to participate, the patient will sign consent forms witnessed by personnel not associated with the study. Patients will be randomized once consent has been obtained.

The patient will then undergo surgery. Operative data will be collected from their chart including implants used, and intraoperative complications. They will be placed in a sling if they are randomized to the sling group and given instructions on passive range of motion exercises to start postoperative day one. If they are assigned to the early motion group they will be placed in a sling for comfort after surgery but told they can remove it when they feel their pain will allow. They will also be instructed on the same passive range of motion program as the sling group. This is different from the standard of care.

Once enrolled, the patients will be randomized through computer randomization then placed in paper packets into either the immobilization group or the early range of motion group.

They will undergo their reverse total shoulder arthroplasty for fracture as they will even if they do not agree to participate in the study (normal treatment)

The immobilization group will be placed in a shoulder abduction sling immediately after surgery for four weeks. They will be allowed to start gentle passive range of motion with forward flexion to 120 degrees, abduction to 90 degrees, and external rotation to 30 degrees. They will receive a home exercise program and formal physical therapy with these limits.

When they come out of the sling at four weeks they will start active range of motion and active assisted range of motion. They cannot internally rotate until 10 weeks after surgery. No formal strengthening until 3 months after surgery.

The early range of motion group will be given a sling for comfort after their surgery. They will be told they can use their arm as tolerated and can remove the sling when comfortable immediately after surgery. They will be allowed to start passive range of motion, active assisted range of motion, and gentle active range of motion with therapy as tolerated with the exception of no internal rotation. They will also not be allowed to strengthen until 12 weeks after surgery. They will get formal physical therapy and be given a home exercise program as well that will be directed by their physical therapist

Both groups will be evaluated postoperatively at 2 weeks, 6 weeks, 12 weeks, 6 months, 1 year, and two years. At each time point the following will be evaluated.

Visual analog pain score American Shoulder and Elbow Society Scores Range of motion Complications Radiographs will be obtained at these visits

Thereported outcome scores will either be recorded in the office or via email using the surgical outcomes system database that is already approved for use at Cooper via legal for quality outcome measures. The patient will be allowed to determine which method they would prefer and is easier for them.

All of these visits will be the same as patients who choose not to enroll in the study. No additional visits are required for the study. The only differences in treatment will be obtaining the patient outcome scores listed above and the random assignment to one of two treatment groups. The random treatment assignments are as follows; the first group of patients will be placed in a sling for four weeks but with early stretching through physical therapy, and the second group will be allowed to use the sling for comfort only and use their arm as tolerated for motion activities such as dressing and bathing. The second group will also receive physical therapy.

The results of the study will not be shared with the subjects or others unless they ask at the completion of the study at which point final data will be revealed to the subjects that ask.

ELIGIBILITY:
Inclusion Criteria:

* Patients 60 years or older who have a displaced proximal humerus fracture
* Meets surgical criteria for a reverse total shoulder arthroplasty
* Receive surgical intervention within 6 weeks of initial injury

Exclusion Criteria:

* Patients <60 years in age
* Patients who cannot undergo surgery due to medical comorbidities
* Patients who receive surgical intervention after 6 weeks from initial injury
* Patients who have preoperative nerve damage from their fractures that would limit the ability to move the arm postoperatively

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients 60 years or older who have a displaced proximal humerus fracture that meet surgical criteria for a reverse total shoulder arthroplasty. Patients are not excluded based on sex
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-02-24 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Early postoperative range of motion | 2 years
  the postoperative range of motion (ROM) will be compared between the 2 groups at 2 weeks, 6 weeks, 12 weeks, 6 months, 1 year, and two years
Postoperative Pain | 2 years
  Patients will rate their pain using the VAS pain scale survey. The visual analog scale (VAS) is a pain rating scale first used by Hayes and Patterson in 1921. Scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm). This scale will be administered to both groups at 2 weeks, 6 weeks, 12 weeks, 6 months, 1 year, and 2 years. The results of these scores will be compared between the two groups at each time point.
Shoulder function | 2 years
  the postoperative shoulder function assessed by the American Shoulder and Elbow Scale (ASES). This scale includes a section on pain (7 items) and a section on activities of daily living (10 items). Scores range from 0 to 100 with a score of 0 indicating a worse shoulder condition and 100 indicating a better shoulder condition. The survey will be administered to both groups at 2 weeks, 6 weeks, 12 weeks, 6 months, 1 year, and 2 years. The results of these scores will be compared between the two groups at each time point.
Postoperative complication | 2 years
  the 2 year postoperative complications will be recorded and compared between the 2 cohorts.
Tuberosity Healing on Radiographs | 2 years
  Radiographic outcomes regarding the degree of tuberosity healing will be obtained at each postoperative visit until the 2 year mark and compared between the 2 cohorts
  After initial imaging, patients will receive subsequent X-rays to monitor tuberosity healing, progression of fracture gap closure with bone formation, and signs of bone resorption. Healing is defined as lack of displacement with consolidation of the fracture and disappearance of previous fracture lines. Displacement will be measured in millimeters compared to position on previous xrays.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine J Fedorka, MD, Principal Investigator — Cooper Hospital Orthopedic Surgery
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hagen MS, Allahabadi S, Zhang AL, Feeley BT, Grace T, Ma CB. A randomized single-blinded trial of early rehabilitation versus immobilization after reverse total shoulder arthroplasty. J Shoulder Elbow Surg. 2020 Mar;29(3):442-450. doi: 10.1016/j.jse.2019.10.005. Epub 2020 Jan 7. PMID 31924519
- [Background] Sheps DM, Silveira A, Beaupre L, Styles-Tripp F, Balyk R, Lalani A, Glasgow R, Bergman J, Bouliane M; Shoulder and Upper Extremity Research Group of Edmonton (SURGE). Early Active Motion Versus Sling Immobilization After Arthroscopic Rotator Cuff Repair: A Randomized Controlled Trial. Arthroscopy. 2019 Mar;35(3):749-760.e2. doi: 10.1016/j.arthro.2018.10.139. PMID 30827428
- [Background] Agorastides I, Sinopidis C, El Meligy M, Yin Q, Brownson P, Frostick SP. Early versus late mobilization after hemiarthroplasty for proximal humeral fractures. J Shoulder Elbow Surg. 2007 May-Jun;16(3 Suppl):S33-8. doi: 10.1016/j.jse.2006.07.004. Epub 2006 Dec 13. PMID 17174113